CLINICAL TRIAL: NCT05613582
Title: The Effectiveness of Transcranial Direct Current Stimulation (tDCS) as Adjunctive Treatment for Chronic Daily Headache in Systemic Lupus Erythematosus: A Double Blind Randomized Multi-Arm Sham Controlled Clinical Trial
Brief Title: The Effectiveness of Transcranial Direct Current Stimulation as Adjunctive Treatment for Chronic Daily Headache in Systemic Lupus Erythematosus
Acronym: SHADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Riwanti Estiasari, MD, PhD, Associate Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22070753
Record Dates: First submitted 2022-10-29; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus; Chronic Headache
Keywords: Systemic Lupus Erythematosus; Chronic Headache; Transcranial Direct Current Stimulation; Double-Blind Study
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Headache Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Primary Motor Cortex (M1) (Experimental): Subjects were randomly assigned to receive tDCS stimulation at the primary motor cortex (M1)
  Interventions: Device: Transcranial Direct Current Stimulation
- Primary Sensory Cortex (S1) (Experimental): Subjects were randomly assigned to receive tDCS stimulation at the primary sensory cortex (S1)
  Interventions: Device: Transcranial Direct Current Stimulation
- Dorsolateral Prefrontal Cortex (DLPFC) (Experimental): Subjects were randomly assigned to receive tDCS stimulation at the dorsolateral prefrontal cortex (DLPFC)
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham (Sham Comparator): The sham intervention procedure was carried out similarly to the experimental group, but in the following group, the device would only conduct electric current in the first and last 30 seconds of the intervention.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — The flow of DC electric current 1 mA for 20 minutes. The position of the electrode placement follows the international EEG 10/20 system.

SUMMARY:
The prevalence of chronic primary headache in Systemic Lupus Erythematosus (SLE) is 54.4%. Several studies have shown that the use of transcranial direct current stimulation (tDCS) at the primary motor cortex (M1), primary sensory cortex (S1), or dorsolateral prefrontal cortex (DLPFC) is effective as adjuvant therapy in primary headache. Using a double-blind design, this clinical trial study will investigate the effectiveness of tDCS as an adjuvant therapy in chronic daily headaches in SLE, by also comparing the effectiveness of administration in the M1, S1, and DLPFC.

The primary endpoint that will be assessed is the frequency of headaches per week, with the secondary endpoints are the degree of headache, quality of life, sleep quality, level of depression, and use of analgesics.

DETAILED DESCRIPTION:
This study aimed to assess the effectiveness of the tDCS protocol as an adjuvant therapy for reducing chronic headache in SLE. It is also hoped that this study will obtain an effective tDCS protocol for chronic headache.

The whole procedure will run for 20 weeks, divided into 3 parts (Pre-intervention, Intervention, and Post-intervention)

Pre-intervention (weeks 0-4) to conduct screening, provide informed consent, and also baseline assessment. Participants will come in weeks 0 and 4.

Intervention (weeks 4-8) to perform the TDCS intervention, record and assess outcomes, and assess if an unwanted event occurs. Participants will come 2 times per week, from week 4 to 8

Post-intervention (weeks 8-20) for continued outcome assessment. Participants will come on weeks 8, 12, 16, and 20

The total number of visits from each participant is 14 times

SLE patients who meet the inclusion criteria and have signed the consent will be subjected to a baseline assessment (weeks 0-4) followed by randomization into 4 groups/arms consisting of 3 treatments (getting standard therapy for SLE and other diseases that have been obtained so far, plus the administration of tDCS at DLPC, M1, S1) and 1 control group that got sham tDCS.

If the tDCS intervention shows effective and safe results, then the subject in the control group (the group that received the sham) will be offered to be given the intervention method at the end of the study.

Any unwanted event (adverse event) that occurs will be recorded. If an undesirable event occurs, a written report will be made to the ethics committee.

Demographic data will be presented descriptively according to the type of data. Normality test will be performed with Shapiro-Wilkins. To find out the changes in the frequency of headaches in the four groups, an analysis using one-way Anova was carried out followed by Bonferroni post hoc analysis with a significance level of 0.05. The effect size of each group will also be analyzed with Cohen's d=02 (small effect), 0.5 (medium) and 0.8 (large) parameters.

Data analysis will be carried out using SPSS 23.0 and GraphPad software.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Patients who have been diagnosed with SLE based on the 2019 ACR criteria
3. Meet the criteria for the diagnosis of chronic headache (criteria based on the International Headache Society, headache occurs in 15 days or more per month, occurs for at least 3 months)

Exclusion Criteria:

1. The patient or the patient's family refuses to participate in the study
2. Is in a state of relapse/flare
3. Allergic reactions / skin infections / wounds / cranial defects / metal implants in the electrode installation area
4. Have a history of brain tumor, severe head injury, stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Headache Frequency | Change from baseline, at the end of weeks 8, and during the follow up period (end of weeks 12, 16, and 20)
  Headache Frequency will be assessed using the headache diary, with a reduced number of frequencies, it indicates a better output

SECONDARY OUTCOMES:
Headache Assessed by Visual Analouge Scale | Change from baseline, 4th, 5th-8th, 12th, 16th, 20th week
  Minimum value: 0 cm Maximum value: 10 cm Assessment using a straight line 10 cm long. Both ends showed signs at 0 cm not painful and the other end at 10 cm very painful. The patient then marks along the line that interprets the pain.
Functional Aspects of Headache-Related Quality of Life Assessed by Chronic Headache Quality of Life Questionnaire (CHQLQ) | 4th, 8th, 12th, 16th, 20th week
  Lowest score 0 Highest score 300 The higher the value, the worse the outcome
Health-Related Quality of Life Assessed by The 36-Item Short Form Health Survey Questionnaire (SF-36) | 4th, 8th, 12th, 16th, 20th week
  Lowest score: 0 Highest score: 100 Higher scores indicate better health status, and a mean score of 50 has been articulated as a normative value for all scales
Sleep Quality Assessed by Pittsburgh Sleep Quality Index (PSQI) | 4th, 8th, 12th, 16th, 20th week
  Lowest score: 0 Highest score: 21 The higher the value, the worse the outcome
Depression level assessed by Mini International Neuropsychiatric Interview Version ICD-10 (MINI ICD 10) | 4th, 8th, 12th, 16th, 20th week
  Will be assessed whether the subject has a depressive episode (Yes/No)
Frequency of use of analgesics | Change from baseline until week 8th, followed at 12th, 16th, 20th week
  Assessment using records of frequency of analgesic consumption
Amount of analgesic use | Change from baseline until week 8th, followed at 12th, 16th, 20th week
  Assessment using records of frequency of amount of analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Riwanti Estiasari, MD, PHD, Principal Investigator — Indonesia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estiasari R, Tiksnadi A, Tunjungsari D, Maharani K, Aninditha T, Sofyan HR, Savitri I, Pangeran D, Jeremia I, Widhani A, Ariane A. Effectiveness of transcranial direct current stimulation (tDCS) as adjunctive treatment for chronic headache in adults with clinically stable systemic lupus erythematosus (SHADE): a randomised double-blind multiarm sham controlled clinical trial. BMJ Open. 2023 Dec 14;13(12):e076713. doi: 10.1136/bmjopen-2023-076713. PMID 38101851